CLINICAL TRIAL: NCT03901859
Title: A Study on the Metabolic Pathway of Tryptophan and Executive Dysfunction in Children With Attention Deficit Hyperactivity Disorder
Brief Title: Metabolic Pathway of Tryptophan and Executive Dysfunction in Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201809043RINA
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2018-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; tryptophan; executive function
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with ADHD: drug-naive patients with ADHD, aged 7-18 year old
- Healthy Controls: drug-naive healthy controls, aged 7-18 year old

SUMMARY:
The present project is to identify the relationship between ADHD and the metabolites of tryptophan.

DETAILED DESCRIPTION:
Because attention deficit hyperactivity disorder (ADHD) is an early onset and long-term impairing disorder with tremendous impact on individuals, families, and societies, detection and diagnosis are very important for ADHD. According to investigators previous work, participants with ADHD have executive dysfunction. Previous studies show that tryptophan is associated with cognitive problems in participants. Analyzing differences in tryptophan metabolites (Indolepropionic acid [IPA], indoleacetic acid [IAA], and kynurenic acid [KYNA]) between participants with ADHD and healthy controls could provide insight into underlying disease pathology of cognitive deficits. In this one-year project, investigators will perform an analysis of tryptophan metabolites in serum to identify potential biomarkers for the executive dysfunction of ADHD.

ELIGIBILITY:
The ADHD group

1. Inclusion Criteria

   Patients with ADHD are eligible to be included in this study only if they meet all of the following criteria:
   1. Patients will be outpatients who are between 7 and 18 years of age.
   2. Patients must have ADHD that meet the Diagnostic and Statistical Manual of Mental disorders, 5th edition (DSM-V) disease diagnostic criteria assessed by the investigator's clinical evaluation, as well as confirmed by the Chinese version of the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Epidemiological Version (K-SADS-E).
   3. Patients must have a Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) score > 4 at baseline.
   4. Patients must be psychotropic drug-naïve. Patients will be considered to be drug-naïve if they have never received medications specifically to treat ADHD.
   5. Patients and parents (or legal representative) must have a degree of understanding sufficient to be able to communicate suitably with the investigator.
   6. Patients must be of normal intelligence in the judgment of the investigator. Normal intelligence is defined as achieving a score of 80 or more when IQ testing is administrated.
   7. Patients must have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests, including neuropsychological testing and venipunctures.
2. Exclusion Criteria

Patients will be excluded from the study if they meet any of the following criteria:

1. Patients with current or past history of schizophrenia, schizoaffective Disorder, organic psychosis, bipolar I or II disorder, autism, or autism spectrum disorder. Other comorbid psychiatric disorders are not excluded if the ADHD symptoms are the primary source of impairment for the patient.
2. Patients with a history of any seizure disorder (other than febrile convulsion) or patients who are taking anticonvulsants for seizure control.
3. Patients have been at serious suicidal risk, determined by the investigator.
4. Patients with a history of alcohol or drug abuse within the past 3 months, or who are currently using alcohol, drugs of abuse, or any described or over-the-counter medication in a manner that the investigator considers indicative of abuse.
5. Patients with cardiovascular disease or other conditions that could be aggravated by an increased heart rate or increased blood pressure.
6. Patients who are likely to need Chinese medicine or health-food supplements that have central nervous system activity.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 120 drug-naïve patients with ADHD, aged 7 to 18 years, will be enrolled. Another 120 healthy participants with matched age and sex will be enrolled in the control group.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Serum level of Indolepropionic acid [IPA] | 1 year
  tryptophan metabolite
Serum level of indoleacetic acid [IAA] | 1 year
  tryptophan metabolite
Serum level of kynurenic acid [KYNA] | 1 year
  tryptophan metabolite

SECONDARY OUTCOMES:
ADHD Rating Scale-IV | 1 year
  behavioral measures
Swanson, Nolan, and Pelham IV scale | 1 year
  The SNAP-IV is a 26-items scale, consisting of the DSM-IV symptoms for the Inattention (Item 1-9) and the Hyperactivity/Impulsivity domains (Item 10-18) of the criteria for ADHD, and the oppositional symptoms (Item 19-26) of the criteria for ODD (20). As in the DSM-IV criteria, to describe psychopathology, the word "often" is included at the beginning of each item, so the precise interpretation of the 4-point rating scale (0 = "not at all", 2 = "just a little", 3 = "quite a bit", and 4 = "very much") reflects the degree that the behavior is abnormally frequent and severe compared to normal childhood behavior.
Achenbach Child Behavior Checklist | 1 year
  designed to assess the competencies and behavioral/emotional problems in children 4-18 for CBCL. rate how true each item is at present or within the last 6 months, using a 3-point response scale. subdivided into a profile report on child's standing in competence items and in 112 problem items. Internalizing score is composed of scores for anxiety/depression, somatic complaints, and withdrawal. Externalizing score is comprised of scores for delinquent behavior and aggressive behavior.
Clinical Global Impressions-ADHD-Severity | 1 year
  The CGI-ADHD-S (120) is a single item clinician rating of the assessment of the global severity of the ADHD symptoms in relation to the clinician's total experience with ADHD patients. Severity is rated on a 7-point scale (1=normal, not at all ill; 7=among the most extremely ill patients). The CGI-ADHD-S will be administered on each visit, from visit 1 through visit 10.
Social Adjustment Inventory for Children and Adolescents | 1 year
  The SAICA is a 77-item semi-structured interview scale that was designed for administration to school-aged children aged 6-18 about themselves, or to their parents about their children (121). The SAICA provides an evaluation of children's current functioning in the domains of (1) school, (2) spare time, (3) peer relations, and (4) home behaviors. A higher mean score (items rated on 4-point Likert scale from 1 to 4) indicates either poorer social function or a more severe social problem (121). (We delete the Spare time relationship in the Overall relationship) The score for each item ranges from 1 to 4. An increased score indicates either a decreased social function or an increased severity of social problem.
Chinese version of the Family Adaptation, Partnership, Growth, Affection, and Resolve | 1 year
  behavioral measures
Cambridge Neuropsychological Test Automated Batteries | 1 year
  neuropsychological measures
Continuous Performance Test | 1 year
  neuropsychological measures

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yung Shang, MDPHD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan